CLINICAL TRIAL: NCT03575247
Title: The Risk of Adrenal Insufficiency and Cushing Syndrome Associated With Glucocorticoid Therapy in People With Chronic Inflammatory Diseases
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Mar Pujades Rodriguez, University Academic Fellow, University of Leeds
Other Study IDs: 16_146
Record Dates: First submitted 2018-06-20; First posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Adrenal; Insufficiency Gluccorticoid-Induced; Cushing; Syndrome or Disease, Glucocorticoid-Induced
MeSH Terms: conditions — Syndrome; Disease | interventions — Glucocorticoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Glucocorticoids — Long-term use of glucocorticoids

SUMMARY:
Glucocorticoids are widely used for the treatment of chronic inflammatory diseases. Although glucocorticoids are effective in controlling disease symptoms, continuous use of the drugs can lead to suppression of adrenal hormones or excessive cortisol level in the blood stream. That is, excess blood cortisol level due to glucocorticoid exogenous supply can either inhibit the 'hypothalamus-pituitary-adrenal axis' for adrenal hormones production or result in Cushing symptoms.

In the period between 1989 and 2008 in the UK, it was estimated that 0.6%-0.8% of the general adult population were long-term users of oral glucocorticoids. However, there is no data on the risk of adrenal suppression and Cushing syndrome due to chronic use of glucocorticoids in the UK to date.

The aim of the study is to investigate the risk of adrenal insufficiency and Cushing syndrome due to long-term use of glucocorticoids in England.

DETAILED DESCRIPTION:
Adrenal insufficiency is a clinical condition that is associated with a deficiency of adrenal hormones, mainly: glucocorticoids and mineralocorticoids. Cushing syndrome is also a condition that stems from the existence of persistent high cortisol level in the body. The majority of Cushing syndrome cases are exogenous (iatrogenic or due to use of medication).

Glucocorticoids are widely used for the treatment of chronic inflammatory diseases. Although glucocorticoids are effective in controlling disease symptoms, continuous use of the drugs can lead to suppression of adrenal hormones or excessive cortisol level in the blood stream. That is, excess blood cortisol level due to glucocorticoid exogenous supply can either inhibit the 'hypothalamus-pituitary-adrenal axis' for adrenal hormones production or result in Cushing symptoms.

In the period between 1989 and 2008 in the UK, it was estimated that 0.6%-0.8% of the general adult population were long-term users of oral glucocorticoids. However, there is no data on the risk of adrenal suppression and Cushing syndrome due to chronic use of glucocorticoids in the UK to date

The aim of the study is to investigate the risk of adrenal insufficiency and Cushing syndrome due to long-term use of glucocorticoids in England. This is a retrospective cohort study of people diagnosed with at least one of six chronic inflammatory diseases (polymialgia rheumatica, giant cell arteritis, systemic lupus erythematosus, rheumatoid arthritis, vasculitis and inflammatory bowel disease).

This study will be based on the analysis of existing primary care health records routinely collected, linked to hospital and mortality data.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old or over
* Registered in a participating general practice for more than 1 year during the study period
* Minimum of 1 year prior to study entry meeting CPRD data quality
* Diagnosed with at least one of the 6 chronic inflammatory diseases

Exclusion Criteria:

* Patients aged under 18 years during the study period
* Registered in general practices that did not consent to data linkage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients registered in CPRD who were eligible for data linkage and had been diagnosed with at least one of six chronic inflammatory diseases (inflammatory bowel diseases, systemic lupus erythematosus, polymyalgia rheumatica, giant cell arteritis, rheumatoid arthritis, and vasculitis) in the period between 1st Jan 1998 and 30th September 2015.
Sampling Method: Non-Probability Sample
Enrollment: 111804 (Actual)
Dates: Start 1998-01-01 (Actual); Primary Completion 2015-01-30 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Glucocorticoid-related adrenal insufficiency | 18 years
  First recorded diagnosis of adrenal insufficiency
Glucocorticoid-related Cushing syndrome | 18 years
  First recorded diagnosis of Cushing syndrome

SECONDARY OUTCOMES:
All cause mortality | 18 years
  Recorded death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Mar Pujades-Rodriguez, PhD, Principal Investigator — University of Leeds

IPD SHARING:
Plan to Share IPD: No